CLINICAL TRIAL: NCT00302744
Title: Effects of Psilocybin in Advanced-Stage Cancer Patients With Anxiety
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center (Other)
Collaborators: Heffter Research Institute (Other)
Responsible Party: Principal Investigator, Charles S. Grob, M.D., professor of psychiatry, Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HEFFTER11287-01
Record Dates: First submitted 2006-03-10; First posted 2006-03-14 (Estimated); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Anxiety
Keywords: Anxiety; Depression; Mood; Cancer; Quality of Life; Psychiatric; Psilocybin; Alternative; Los Angeles
MeSH Terms: conditions — Anxiety Disorders; Depression; Neoplasms | interventions — Psilocybin; Pharmaceutical Preparations; Niacin; Niacinamide

STUDY DESIGN:
Intervention Model Description: Within-subject cross-over study. Each participant received active drug and active placebo on separate dates.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Psilocybin (Experimental): Single, 6-hour treatment with 0.2 mg/kg active psilocybin capsule.
  Interventions: Drug: Psilocybin (drug); Diagnostic Test: MRI
- Active Niacin Placebo (Active Comparator): Each subject functioned as their own control, receiving niacin placebo capsule in a single 6-hour session.
  Interventions: Other: Niacin; Diagnostic Test: MRI

INTERVENTIONS:
Drug: Psilocybin (drug) — Capsule (.2 mg/kg).
  Other Names: 4-phosphoryloxy-N,N-dimethyltryptamine
  Arms: Psilocybin
Other: Niacin — Active Placebo
  Other Names: nicotinamide; vitamin B3
  Arms: Active Niacin Placebo
Diagnostic Test: MRI — MRI required for study inclusion for purpose of ruling out metasteses to brain

SUMMARY:
Psychiatric Research Study For Cancer Patients

The Los Angeles Biomedical Research Institute at Harbor-UCLA Medical Center is conducting a study designed to measure the effectiveness of the novel psychoactive medication psilocybin on the reduction of anxiety, depression, and physical pain.

DETAILED DESCRIPTION:
The significance of this study is that it is addressing the important issues of psychological and spiritual well being of people who have advanced cancer. In 2001, the National Cancer Policy Board of the Institute of Medicine and National Research Council issued a report (Improving Palliative Care for Cancer: Summary and Recommendations) that specifically recommended research be conducted using novel agents and methods. Psilocybin is a novel agent which produces a profound alteration in your state of consciousness. It is the main active ingredient found in "magic mushrooms".

Our specific aim is to learn whether this psychoactive drug, psilocybin, might be effective in reducing anxiety, depression and physical pain, and therefore improving your quality of life. This pilot study will start with 12 people ages 18-70. For each participant there will be two overnight admissions to the hospital. In one session you will be given a placebo and in the other you will get the active medication, but no one will know which drug is administered when. This is called a double blind study. You will be asked to fill out questionnaires about how you feel, your pain levels and your moods. There will also be at least two psychotherapy meetings before the study sessions, so that you are fully aware of what to expect and to have all your questions answered.

We cannot take you in the study if you have central nervous system (CNS) cancers, kidney disease, diabetes, abnormal liver function tests, epilepsy, cardiovascular disease including untreated high blood pressure (BP greater than 140/90), and pregnancy. The psychiatric exclusions are: you or an immediate family member with a history of a major psychiatric disorder, a current substance abuse problem, or an anxiety or a mood disorder within 1 year prior to the onset of symptoms of your current illness.

We also cannot take you in the study if you are taking certain medications, such as: anti-seizure, insulin and oral hypoglycemics, and cardiovascular drugs (except anti-hypertensive medications). Some antidepressant (SSRIs) medications cannot be taken within the two weeks prior to the session (except for Prozac, which cannot be taken in the last 5 weeks prior to the session).

You will get a MRI of the brain prior to admission (if you haven't had one in the prior two months), at the study's expense, to be sure there is no CNS involvement. You can provide us, or the study will pay for, lab work from the prior 2 weeks (CBC, liver function and renal function). The history and physical, neurological exam, EKG, and a urine pregnancy test (if you are a woman with child-bearing potential), will be done on admission by the house staff doctors.

You will be allowed to take your own medications while in the hospital, and will be encouraged to bring to the hospital personal photos, small memorabilia, and some of your favorite music that can be played during the sessions.

ELIGIBILITY:
Inclusion Criteria:

* Have advanced-stage cancer and anxiety.
* Be between the ages of 18 - 70.

Note: The location for the two treatment sessions is Los Angeles, California. Treatment sessions are scheduled three to six weeks apart, and they include one overnight hospital stay both times.

Exclusion Criteria:

* Not have cancer that affects the central nervous system or brain function.
* Have no history of major psychiatric disorder.
* Have no kidney disease, abnormal liver functions, epilepsy, or cardiovascular disease, including untreated hypertension.
* Not be taking insulin, oral hypoglycemic, anti-seizure, or cardiovascular medications (except anti-hypertensive drugs).
* May take PRN benzodiazepines up to 3 days before the session.
* No Prozac for the previous 5 weeks.
* No medications the day of and the day after treatment sessions, except may take ongoing adjuvant chemotherapy as prescribed, prescribed or over-the-counter non-narcotic pain medication at any time, and narcotic pain medications up to eight hours before administration of psilocybin and six hours after administration.
* No alcohol consumption the day before, the day of, and the day after a session.
* Female subjects of childbearing potential must have a negative pregnancy test and agree to use an effective form of birth control.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2004-04; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Anxiety | 6 months
  State-Trait Anxiety Inventory for Adults - Form Y-2

CONTACTS AND LOCATIONS:
Overall Officials: Charles S. Grob, MD, Principal Investigator — University of California, Los Angeles
Locations (1):
- Harbor-UCLA Medical Center, Torrance, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Grob CS, Danforth AL, Chopra GS, Hagerty M, McKay CR, Halberstadt AL, Greer GR. Pilot study of psilocybin treatment for anxiety in patients with advanced-stage cancer. Arch Gen Psychiatry. 2011 Jan;68(1):71-8. doi: 10.1001/archgenpsychiatry.2010.116. Epub 2010 Sep 6. PMID 20819978